CLINICAL TRIAL: NCT07027865
Title: Targeting Added Sugar to Improve Dietary Intake in High-risk Adolescents
Brief Title: Sip and Snack Better (SSB) Study: Improving Added Sugar in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 28611; K01HL153783 (NIH); R03HL171171 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-06-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Dietary Habits; Diet, Healthy
Keywords: dietary intake; added sugar; adolescents; behavior change; dietary intake assessment
MeSH Terms: conditions — Feeding Behavior | interventions — RBM14 protein, human; SSB protein, human; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching Behavioral Intervention (Experimental): Behavioral intervention using health coaching and technology to improve dietary intake
  Interventions: Behavioral: Sip & Snack Better (SSB) Intervention
- Technology-Only Comparison (Other): Digitally-delivered nutrition education only comparison arm
  Interventions: Other: Sip & Snack Better (SSB) Tech-Only Comparison

INTERVENTIONS:
Behavioral: Sip & Snack Better (SSB) Intervention — Participants (teens 12-16 years) and their parent or legal guardian will participate in a 12-week health coaching intervention to reduce added sugar intake. Parents and teens will participate in 6 health coaching sessions (in weeks 1, 3, 5, 7, 9, and 12; 30-45 minutes, online via Zoom). Teens will participate in four in-person groups sessions (in weeks 2, 4, 6, and 8) and receive text-messages to reinforce intervention content.
  Arms: Health Coaching Behavioral Intervention
Other: Sip & Snack Better (SSB) Tech-Only Comparison — Participants (teens 12-16 years) and their parent or legal guardian will participate in a 12-week technology-only comparison arm. Parents and teens will receive information about added sugar intake and healthy eating once via email or text message (based on preference) in weeks 1, 3, 5, 7, 9, and 12. Teens will receive informational text messages 3 times per week .
  Arms: Technology-Only Comparison

SUMMARY:
Teens consume more added sugar than any other age group. Too much added sugar is associated with poor diet quality, obesity risk, and negative cardiometabolic outcomes. Behavioral interventions to improve dietary intake are needed, but are currently lacking for this age group. This study aims to test how feasible, acceptable, and effective a 12-week contextually-tailored health coaching program, called Sip & Snack Better (SSB), is in reducing added sugar in teens, compared to a technology-only comparison. It will provide important information on how to improve dietary intake and reduce added sugar in teens. Additionally, measuring diet is very challenging in teens, so this study will also test the use of an objective biomarker (called the carbon isotope ratio (CIR)) as a measure of added sugar intake before, during, and after the 12-week study.

ELIGIBILITY:
Inclusion Criteria:

* Parent is 18 years or older, and the legal guardian of the adolescent
* Adolescent is between the ages of 12 and 16 years
* Parents and adolescents have the ability to read, write, and understand English
* Adolescents have a cell phone and are willing to use it to receive text messages and answer survey questions
* Parents and adolescents live in the Philadelphia region and can attend in-person visits at the research center in North Philadelphia
* Parents and adolescents can access video communication platforms (i.e., Zoom) via phone or computer
* Parents and adolescents are willing to be randomized to either treatment condition
* Adolescents exceed daily recommendations for added sugar intake (as assessed by dietary screener)

Exclusion Criteria:

* Adolescent has a medical condition that influences weight status or added sugar intake (e.g., Type 1 or Type 2 diabetes)
* Adolescent has a psychological or psychiatric condition that prevents study participation without individualized support (e.g., autism spectrum disorder)
* Adolescent has been diagnosed with or has received/is receiving treatment for an eating disorder
* Adolescent has been diagnosed with or has received/is receiving treatment for depression
* Adolescent has dietary restrictions, dietary prescriptions, or dietary goals given by a health care provider that would influence weight or added sugar intake

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Added Sugar Intake | Baseline to 12-weeks
  Change in added sugar intake will be assessed using the carbon isotope ratio (CIR) as a objective measure of added sugar intake via breath, blood, and hair samples taken at baseline and post-intervention. Intent-to-treat analyses will be conducted using linear regression models to examine changes in CIR between intervention and control participants. A lower (i.e., more negative) CIR value indicates lower added sugar intake.
Intervention Feasibility | Baseline to 12-weeks
  Feasibility will be assessed by session attendance (>75%) and retention (>80%) over the 12-week study.
Intervention Acceptability | Baseline to 12-weeks
  Participants will report acceptability (>80% rating of 4 or 5 on Likert scale questions) on a post-intervention acceptability questionnaire

SECONDARY OUTCOMES:
Changes in Diet Quality | Baseline to 12-weeks
  Changes in diet quality will be assessed via Healthy Eating Index (HEI) derived from three 24-hour dietary recalls at baseline and post-intervention. HEI is scored on a scale from 0 to 100 with higher scores indicating higher diet quality.

OTHER OUTCOMES:
Feasibility of Breath CIR | Baseline to 12-weeks
  Feasibility of breath CIR to capture intervention adherence will be assessed via completion rates of breath samples (>80%). The sampling protocol collects three breath samples on five random sampling days at baseline and in weeks 3, 6, 9, and 12 (15 total breath samples over 12-weeks).
Predictive Accuracy of the Carbon Isotope Ratio (CIR) as an indicator of Added Sugar and Sugar Sweetened Beverage Intake | Baseline to 12-weeks
  Area under the curve (AUC) models will be used to determine how well each CIR sample type (blood, breath, hair, nails) captured changes in added sugar and sugar-sweetened beverage intake (derived from 24-hour dietary recalls). AUC ranges from 0 -1 and a higher AUC indicates better model fit.
CIR Biomarker Acceptability | Baseline to 12-weeks
  Participants will report on a scale of 1-5 how anxious or stressed they are before the collection (1= Very stressed or anxious, 5= Not at all stressed or anxious). After collection, participants will report on a scale of 1-5 how comfortable they felt during the collection (1= very uncomfortable, 5= very comfortable) and how difficult or burdensome they found the collection method (1=very difficult or very burdensome, 5=not at all difficult or burdensome). After all data are collected participants will rank the collection methods in order of preference (1= top choice, 4= last choice) and report (yes/no) if they would be willing to provide each type again in a subsequent study (breath, blood, hair, nail).

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Obesity Research and Education, Philadelphia, Pennsylvania, United States